CLINICAL TRIAL: NCT01631682
Title: Psychophysiology of Delayed Extinction and Reconsolidation in Humans
Brief Title: Pilot Study of Pharmaceutical and Behavioral Interventions to Treat Anxiety Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott Orr, Associate Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: W81XWH-11-2-0092
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Posttraumatic Stress Disorder; Anxiety Disorder
Keywords: Posttraumatic Stress Disorder; PTSD; Anxiety; Fear of spiders; Reconsolidation; Reconsolidation blockade
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Arachnophobia | interventions — Propranolol; Mifepristone; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Propranolol (Active Comparator): a single dose of 40mg propranolol may be given to begin visit 2, followed by 90min wait and subsequently CS reactivation
  Interventions: Drug: Propranolol
- Reactivation with time delay (Active Comparator): For those not receiving propranolol on visit 2, one experimental CS will be reactivated, followed by a 10 minute break and subsequently extinction
  Interventions: Behavioral: Reactivation
- Mifepristone (Experimental): a single dose of 1800mg (200mg tablets) mifepristone may be given to begin visit 2, followed by 90min wait and subsequently CS reactivation
  Interventions: Drug: Mifepristone
- Intranasal oxytocin (Experimental): A single 32IU dose of Syntocinon (intranasal oxytocin) is given to begin visit 2, followed by a 10 minute wait and subsequent CS reactivation.
  Interventions: Drug: Intranasal oxytocin

INTERVENTIONS:
Drug: Propranolol — 40mg single pill
  Other Names: Inderal
  Arms: Propranolol
Behavioral: Reactivation — subject is re-exposed to CS+R on day 2 (code for CS that is both paired with shock and reactivated on day 2)
  Arms: Reactivation with time delay
Drug: Mifepristone — 1800mg, 9 tablets
  Other Names: Mifeprex; Korlym
  Arms: Mifepristone
Drug: Intranasal oxytocin — 32 IU, 8 self-administered intranasal sprays, 4 in each nostril
  Other Names: Syntocinon
  Arms: Intranasal oxytocin

SUMMARY:
The aim of this project is to create fear conditioning paradigm within which the relative strengths of various novel pharmacological and behavioral interventions can be tested. These interventions are intended to reduce the fearfulness associated with fear conditioning by blocking a memory process known as reconsolidation. In fear conditioning, a "conditioned" stimulus (CS) is paired with an aversive "unconditioned" stimulus (US) such as an electric shock, until presentation of the CS alone comes to elicit a fear conditioned response (CR). The investigators hypothesize that by using a more highly prepared CS (i.e. video of spiders); more sensitive subjects (individuals with stronger acquired CRs); and additional experimental probes for the presence of the latent CR, the investigators may develop a normal human paradigm that is not plagued by previously observed floor effects (i.e. intervention is 100% effective), within which both the established techniques of propranolol and delayed extinction will produce significant, but only partial, CR reduction. This would leave room to test and compare potentially more powerful candidate reconsolidation-blocking or memory-updating interventions. To achieve these aims, subjects will undergo a four-day fear conditioning and delayed extinction protocol. Skin conductance response data will be gathered across the different phases of the experiment.

DETAILED DESCRIPTION:
1. BACKGROUND AND SIGNIFICANCE 1.1. Reconsolidation and its modification. Recent animal research suggests that reactivation (retrieval) of a consolidated memory can return it to a labile state from which it must be restabilized in order to persist. This stabilization process has been termed "reconsolidation," and various behavioral and pharmacologic interventions have been found to modify or block it. Although extinction can reduce or even apparently eliminate conditioned fear, it typically does so by inhibiting the expression of the fear memory, not by erasing it. In contrast, blockade of reconsolidation is believed to erase, or at least diminish, the fear memory trace. It is not uncommon for reconsolidation articles to conclude with a statement that this offers novel therapeutic possibilities for PTSD, which may in part be characterized as a disorder of over-consolidated, persistently disturbing memories that do not go away.1
2. SPECIFIC AIM The aim of this project is to create an experimental assay in the form of an optimal Pavlovian differential fear conditioning paradigm, within which the relative strengths of various novel pharmacological and behavioral, reconsolidation-blocking interventions can be tested. As impressive as the Kindt8 and Schiller10 studies are for demonstrating pharmacological and behavioral fear reconsolidation-blocking interventions in normal humans, the results produced by these interventions make them nearly useless as potential assays for reconsolidation blockade. Specifically, both interventions produced an apparent total abolition of the fear memory, i.e., they both contain a floor effect. The aim in this work is to develop a normal human paradigm within which both propranolol and delayed extinction produce significant, but only partial reduction of the CR, which might then be improved upon by more powerful reconsolidation-blocking interventions. This study will not be used to support a label, advertising, or indication change of propanolol, and will not be prescribed in a patient population, route of administration, or dosage that significantly increases risk.

   2.1. Elements of a new design to eliminate the floor effect 2.1.1. A stronger US. One way to produce a CR that is more resistant to reconsolidation blockade, i.e., to reduce the floor effect, would be to use a stronger US. However, because in our ongoing human conditioning studies, we are already using an electric shock selected in advance by subjects to be "highly annoying but not painful," we believe that to use a level of shock above this would be ethically impermissible, and hence we will not pursue this possibility.

   2.1.2. A more highly "prepared" CS. It has long been shown that certain classes of CSs, when paired with a US, produce a stronger fear CR, i.e., they are more "prepared" to enter into an association with the US.13 The Schiller design10 did not use a prepared CS, but the Kindt study8 did, viz., still pictures of spiders. In our design, we will enhance the preparedness of the CS by using 12-sec.14 high-definition video clips of three different crawling tarantulas, each conspicuously different in appearance. Importantly, however, the present project will not be a study of spider fear or phobia; we will only use high-definition videoto enhance CS preparedness.

   2.1.3. More sensitive subjects. We will limit recruitment to subject candidates who fall within the upper half of the distribution of normal humans on the Spider Phobia Questionnaire-1515 (SPQ-15) and for whom the CSs are likely to be especially salient. However in order to avoid potential adverse clinical consequences of participation, we will exclude subjects with features of diagnosable spider phobia (or the presence of any other Axis I mental disorder).

   2.1.4. Selecting subjects with stronger CRs. In order for a subject who has completed the Day 1 Acquisition phase of the experiment to proceed to the remaining phases, we will require that they show strong evidence of conditioning, as manifest in CRs greater than 0.25 µSiemens to at least two CS+s. The Schiller study10 employed a differential conditioning cut-off of 0.10 µSiemens, but based upon our own experience, we favor the raw score cut-off. The Kindt study8 employed no such cut-off.

   2.1.5. Employing additional probes for the presence of the latent CR. The Kindt8 and Schiller10 studies employed two of the four available techniques for revealing the presence of the latent CR: spontaneous recovery and reinstatement. In the present experiments, we will also examine renewal and savings. These will require that the CSs be presented in different contexts, which will be achieved in the following manner. Each of the three different tarantulas will appear within three different backgrounds, or contexts, resulting in a 3 x 3 design, and a total of nine different video clips. The use of high-definition video on a large-screen television will help to reduce the context-with-a-context problem. The sequence of presentation of the nine clips will be pseudorandomly varied across subjects within a group, and identical across groups.
3. SUBJECT SELECTION 3.1. Inclusion/Exclusion Criteria 3.1.1. Inclusion criteria. 1) Age 18-35 2) Top half of the normal human distribution of the Spider Phobia Questionnaire-15.

   3.2. Exclusion criteria 3.2.1. Exclusion criteria prior to undergoing first experimental session. 1) Any of the following criteria for diagnosable spider phobia: a) marked or persistent fear of spiders that is excessive or unreasonable; b) intense anxiety or panic upon exposure to a spider; c) avoidance of spiders, anxious anticipation of exposure to spiders, or distress in the presence of spiders, any of which interferes significantly with the person's normal routine, occupational or academic functioning, or social activities or relationships; or d) marked distress about having fear of spiders; 2) Any current Axis I mental disorder on the Structured Clinical Interview for DSM-IV (SCID); or 3) presence of drugs of abuse, e.g., opiates, marijuana, cocaine, or amphetamines, as determined by urine testing. Additionally (4) non-English-speaking subject candidates will be excluded because validated versions of some of the instruments and questionnaires to be administered are not available in other languages.

   3.3. Recruitment methods. Healthy subject candidates will be drawn from advertisements in the media. Most subject volunteers are expected to be drawn from the pool of 250,000 students in the Boston area. No employees or students supervised by the Investigators will be enrolled in this study, nor will Harvard Medical School students. Candidates who express an interest in participating will be scheduled to make a visit to our laboratory for an evaluation as to whether they satisfy the inclusion and exclusion criteria.
4. SUBJECT ENROLLMENT Prior to the initiation of the study procedures, an investigator will obtain the written informed consent using the form approved by the Partners Human Research Committee. If drugs are potentially involved, this will be a licensed physician investigator.
5. STUDY PROCEDURES 5.1. Design. We will use SCR as the measure of the CR. We have chosen SCR because we have 25 years' experience with this dependent measure in human conditioning studies.20 Intertrial intervals will vary within 15 and 25 sec. with a mean of 20 sec. Two active reconsolidation-blocking interventions will be employed: 1) Propranolol reactivation as in Kindt,8 and 2) Reactivation-delayed extinction as in Schiller.10 Subjects will be randomized to one of three conditions: propranolol (40mg; single dose); placebo (single dose); behavioral (no pill). The research pharmacy will create and manage the randomization list. The study will be single blind. The experimental phases will comprise three consecutive days and a fourth day one month later. Prior to beginning the experiment, the subject will set their own level of electric stimulation (shock). They will be instructed to choose a level that is highly annoying but not painful. The experimenter will start the stimulation at a very low, nearly imperceptible level and gradually increase the level until the subject says "stop." That level will then be used throughout the experimental sessions.

   5.1.1 Day 1 5.1.1.1 Interview and Questionnaire. Candidates for this project will undergo a comprehensive evaluation to assess psychiatric and medical history and a structured clinical interview to confirm lack of psychiatric diagnoses (SCID). Subjects will also complete the SPQ-15.15 Eligible candidates will proceed to Habituation and Acquisition.

   5.1.1.2 Habituation and Acquisition. Subjects will view video of three rooms (contexts), different in color and content, presented on a 42" high definition television. The conditioned stimuli (CSs) will be three different videos of tarantulas, one presented in each room. Two of the three tarantulas will serve as the two CS+s and the third as the CS-. Each CS+ presentation will sometimes be followed by shock (i.e., reinforced); the CS- will never be followed by shock. Day 1 will consist of two sequential components: a) 2 unreinforced presentations of each CS (habituation), followed by b) 8 presentations of each CS, with 5 of each CS+ presentations followed by shock (i.e., 63% reinforcement, acquisition). All Day 1 CS presentations will occur within Context A.

   5.1.2. Day 2 (Intervention) will consist of either 1) propranolol (40 mg oral) or placebo (oral) followed 90 min. later by a single, unreinforced presentation of one of the two CS+s, designated the reactivated CS+ (CS+R) (after Kindt8); or 2) a single, unreinforced presentation of the CS+R without receiving a pill, followed 10 min. later by a) 10 further unreinforced CS+R presentations; b) 11 unreinforced presentations of the remaining CS+, designated the CS+ with no intervention (CS+N); and c) 11 CS- presentations (after Schiller10). Subjects will be randomized to one of these three interventions (propranolol, placebo, or behavioral) following Day 1. All Day 2 CS presentations will take place within Context B.

   5.1.3. Day 3 (Renewal, Reinstatement) will consist of three sequential components: a) 2 unreinforced presentations each of the CS+R, CS+N, and CS- (renewal test trials); b) 3 presentations of the US alone, and c) 8 further unreinforced presentations each the CS+R, CS+N, and CS- (reinstatement test trials, also re-extinction). All Day 3 CS presentations will occur within Context A.

   5.1.4. Day 30 (Spontaneous Recovery/Renewal, Savings) will consist of two sequential components: a) 8 unreinforced presentations each of the CS+R, CS+N, and CS- (spontaneous recovery test trials, also re-extinction); and b) 8 presentations each of the two CS+s with 63% reinforcement, and the CS- (savings test trials during re-acquisition). All Day 30 CS presentations will occur within Context C.

   The following numbers of shocks will be delivered to each subject: Day 1: 10 shocks, Day 2: 0 shocks, Day 3: 3 shocks, Day 30: 10 shocks.
6. BIOSTATISTICAL ANALYSIS 6.1. Statistical approach. Data from the above experiments will be subjected to analysis of variance techniques similar to those fully described in the Kindt article8 and supplement, Schiller article10 and supplement, as well as in our published human differential conditioning studies.14,16-19

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Top half of the normal human distribution of the Spider Phobia Questionnaire-15

Exclusion Criteria:'

* Any criteria for diagnosable spider phobia
* Any current Axis I mental disorder on the Structured Clinical Interview for DSM-IV (SCID)
* Presence of drugs of abuse (e.g. opiates, marijuana, cocaine, or amphetamines) per urine screen
* Non-English speaking (due to lack of validated questionnaires/instruments in other languages)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2010-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott P. Orr, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- [Result] Fricchione J, Greenberg MS, Spring J, Wood N, Mueller-Pfeiffer C, Milad MR, Pitman RK, Orr SP. Delayed extinction fails to reduce skin conductance reactivity to fear-conditioned stimuli. Psychophysiology. 2016 Sep;53(9):1343-51. doi: 10.1111/psyp.12687. Epub 2016 Jun 17. PMID 27314560
- [Result] Spring JD, Wood NE, Mueller-Pfeiffer C, Milad MR, Pitman RK, Orr SP. Prereactivation propranolol fails to reduce skin conductance reactivity to prepared fear-conditioned stimuli. Psychophysiology. 2015 Mar;52(3):407-15. doi: 10.1111/psyp.12326. Epub 2014 Sep 16. PMID 25224026

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 186 individuals initially signed a consent form. Of these 186 individuals who gave signed consent, 14 had unmeasureable skin conductance levels and were not able to participate in the study, leaving 172 individuals who participated.
Groups:
- Reactivation With Time Delay: For those not receiving propranolol on visit 2, one experimental CS will be reactivated, followed by a 10-min break and then extinction.
  Subject is re-exposed to CS+R on day 2 (code for CS that is both paired with shock and reactivated on day 2)
Period: Overall Study
Arm/Group | Propranolol | Reactivation With Time Delay | Mifepristone | Intranasal Oxytocin
Started | 55 | 66 | 44 | 7
Completed | 24 | 21 | 13 | 5
Not Completed | 31 | 45 | 31 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Reactivation With Time Delay | Mifepristone | Intranasal Oxytocin | Total
Number analyzed (Participants) | 24 | 21 | 13 | 5 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 13 | 5 | 63
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (3.2) | 23.1 (2.6) | 23.2 (4.5) | 22.8 (3.3) | 22.9 (3.4)
Gender [Count of Participants; unit: Participants]
  Female | 12 | 10 | 7 | 5 | 34
  Male | 12 | 11 | 6 | 0 | 29
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 13 | 5 | 63
Spider Phobia Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Range of scores = 0-15. Higher score represents greater fear of spiders.
  units on a scale | 8.0 (1.8) | 7.6 (2.0) | 8.0 (2.5) | 7.0 (2.6) | 7.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Skin Conductance Response
Description: Skin conductance response (SCR) is the change in skin conductance level in response to a stimulus. We compared the SCR to a non-treated conditioned stimulus (CS+N) with the SCR to a treated conditioned stimulus (CS+R) by creating a difference score (CS+R - CS+N) for the day 3 data. Day 3 is 48 hours after the fear-conditioning procedure and serves as the primary measure of whether the treatment had an effect. SCR was measured in microSiemens; the SCR difference score reflects a change in microSiemens.
Time Frame: 48hrs
Measure: Mean (Standard Deviation); unit: microSiemens
Arm/Group | Propranolol | Reactivation With Time Delay | Mifepristone | Intranasal Oxytocin
Number analyzed (Participants) | 24 | 21 | 13 | 5
microSiemens | .06 (.34) | .17 (.44) | -1.27 (1.68) | -.04 (.27)
Statistical Analysis 1: Comparison: Propranolol; This study used a within-groups design. Each subject provides his/her own comparison data. It was predicted that that a conditioned stimulus that was reactivated (CS+R) after propranolol was administered would result in a smaller SCR than a conditioned stimulus that was not reactivated (CS+N); Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 2: Comparison: Reactivation With Time Delay; This study used a within-groups design. Each subject provides his/her own comparison data. It was predicted that that a conditioned stimulus that was initially presented (CS+R) and then followed by a series of extinction trials after a 10-min delay would result in a smaller SCR than a conditioned stimulus (CS+N) that was not extinguished without a 10-min delay; Test type: Superiority or Other; p > .05, ANOVA
Statistical Analysis 3: Comparison: Mifepristone; This study used a within-groups design. Each subject provides his/her own comparison data. It was predicted that that a conditioned stimulus that was reactivated (CS+R) after mifepristone was administered would result in a smaller SCR than a conditioned stimulus that was not reactivated (CS+N); Test type: Superiority or Other; p < .05, ANOVA
Statistical Analysis 4: Comparison: Intranasal Oxytocin; This study used a within-groups design. Each subject provides his/her own comparison data. It was predicted that that a conditioned stimulus that was reactivated (CS+R) after intranasal oxytocin was administered would result in a smaller SCR than a conditioned stimulus that was not reactivated (CS+N); Test type: Superiority or Other; p > .05, ANOVA

ADVERSE EVENTS:
Time Frame: Within 24 hours.
Arm/Group | Propranolol | Reactivation With Time Delay | Mifepristone | Intranasal Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/13 | 0/5
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 2/13 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propranolol (N=24) | Reactivation With Time Delay (N=21) | Mifepristone (N=13) | Intranasal Oxytocin (N=5)
Mild Nausea (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Mild nausea, possibly related to the medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes